CLINICAL TRIAL: NCT02331017
Title: Assessment of the Contribution of the Combined Acoustic Hearing Via a Hearing Aid and Electric Hearing Via a Cochlear Implant in Adult Bimodal Users With Moderate to Severe Residual Hearing in the Implanted and Non Implanted Ear.
Brief Title: Assessment of Bimodal Contribution in Adult Cochlear Implant Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, MICHAL.LUNTZ, Head of the Otolaryngology Head and Neck Surgery Department, Bnai Zion Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BZ0084
Record Dates: First submitted 2014-12-24; First posted 2015-01-05 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Deafness
Keywords: Bimodal; Cochlear Implant; Hearing aid; Auditory Perception
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bimodal users (Experimental): Bilateral-bimodal users with moderate-to-severe hearing loss who use hearing aids for at least 75% of their waking hours.
  Administration of Speech perception tests and self-rating questionnaire
  Interventions: Behavioral: Speech perception tests and self-rating questionnaire

INTERVENTIONS:
Behavioral: Speech perception tests and self-rating questionnaire — Speech perception test results and self-rating questionnaire scores will be analyzed by means of non-parametric statistical tests. The statistical tests will be chosen in accordance with the number and type of variables in each test. Correlation between audiological variables (aided and unaided hearing thresholds in the non implanted ear, aided speech perception abilities in the HA-alone condition) and the bilateral-bimodal benefit will be examined. Moreover, possible relationship between self-rating questionnaire scores and speech perception test results will be assessed.

SUMMARY:
To evaluate the combination of electric hearing through Cochlear Implant and acoustic hearing through hearing aid in bimodal users with moderate-to-severe hearing loss in the non-implanted ear. The research will also provide pilot study data on unilateral Cochlear Implant recipients with residual useful acoustic hearing in the implanted ear whose acoustic hearing has been preserved.

DETAILED DESCRIPTION:
Many current unilateral Cochlear Implant users have some residual acoustic hearing in the opposite ear as well as in the implanted ear. The amount of useful residual acoustic hearing varies among these implantees. There are several acoustic and electric combinations in the bilateral-bimodal listening mode depending on the amount of useful residual acoustic hearing in each ear. The combination of low frequency acoustic information provided by the hearing aid on each ear, completes the high frequency electric information provided by the Cochlear Implant (complementary bimodal benefit). Each of the different rehabilitation combinationsfor unilateral Cochlear Implant users enablesa unique integration of the three aspects of bilateral hearing bilaterality, binaurality and bimodality which may provide significant advantages over unilateral Cochlear Implant stimulation in terms of speech perception in noise, complementary information as well as localization abilities.

The study will include 20 bilateral-bimodal users with moderate-to-severe hearing loss at 250 Hz, 500 Hz and 1000 Hz in the non-implanted ear, who use hearing aids for at least 75% of their waking hours. Evaluation utilizes bilateral-binaural and bimodal complementary effects task-specific test batteries based on published doctoral research project. The assessment protocol consisted of tests that include various speech materials, different maskers, presentation of the noise from different locations in space, right/left speech lateralization, pitch-related tasks and subjective questionnaires. All tests will be administered in three listening conditions: Cochlear Implant -alone, hearing aid-alone and Cochlear Implant +hearing aid.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral-bimodal users
* With moderate-to-severe hearing loss at 250 Hz, 500 Hz and 1000 Hz in the non-implanted ear
* Who use hearing aids for at least 75% of their waking hours

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Speech perception task specific tests using assessment protocol which will include 6 speech perception tests in quiet and noise listening conditions. | 12 months
  ests designed to examine the contribution of bilateral-binaural benefits:
  1. Semantically unpredictable sentence recognition presented from the front in the presence of a two-male-talker masker.
  2. Horizontal right/left speech lateralization in quiet
  3. Perception of monosyllabic words (HAB) in competing three-male-talker babble.
  4. Semantically unpredictable sentence recognition in the presence of one competing talker using a reversed speech sentence spoken by only two different talkers with different F0 characteristics.
  5. Perception of intonation.
  6. Evaluation of the difference between the perception of natural prosody speech and the perception of speech with flattened F0 contour

SECONDARY OUTCOMES:
Assessment of functional performance in daily life using self-repot questionnaires | 12 months
  the Speech, Spatial and Quality (SSQ) questionnaire and the Hearing Handicap Questionnaire (HHQ).
Standard basic speech perception tests | 12 Months
  Standard basic speech perception tests which will enable to characterize the basic speech perception abilities of the bilateral-bimodal users by means of a commonly utilized assessment tool: monosyllabic word discrimination on the Hebrew version of the AB Word List (HAB) in quiet; Hebrew version of the CID sentence recognition test in quiet and the Hebrew version of the CID sentence recognition test in the presence of four-talker-babble noise with the SNR fixed at +5dB, speech and noise presented from the front.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Luntz, MD, Principal Investigator — Bnai Zion Medica Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel